CLINICAL TRIAL: NCT03343821
Title: Analysis of the French Balance and Daily Life (EVQ) Questionnaire for Evaluation of Balance in the Frail Elderly
Acronym: EVQ
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2016/CEDMH-02; 2017-A01007-46 (Other: ANSM)
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2019-08

CONDITIONS: Accidental Fall

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Frail elderly patient
  Interventions: Other: Balance and daily life questionnaire

INTERVENTIONS:
Other: Balance and daily life questionnaire — Patients complete questionnaire

SUMMARY:
The Balance and Daily Life questionnaire (EVQ) observes the adaption of the patient in six scenarios of daily life; it is a measurement of falls, but also an evaluation of the modifications taken to prevent future falls. This study will analyze the robustness of this questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient is at least 65 years' old
* The patient is fragile (< 8 score ≤ 11 SEGA score) hospitalized in the Physical Medicine and Functional Geriatric Readaptation service of the CHU Nîmes
* The patient can walk autonomously for 20m (with or without a walking aid)
* The patient is allowed to weight-bear

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent form
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* The patient is forbidden to weight-bear
* Comprehension problems preventing the accomplishment of the tasks
* Major short-term memory problems preventing the accomplishment of the tasks

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: • Frail elderly patients over 65 years old hospitalized in the Physical Medicine and Functional Geriatric Readaptation service of the CHU Nîmes
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
Inter-evaluator reliability of Balance and Daily Life Questionnaire | Day 0
  Balance and Daily Life Questionnaire assessed by 2 evaluators
Temporal stability of Balance and Daily Life Questionnaire | Day 3
  Balance and Daily Life Questionnaire given 3 days apart

SECONDARY OUTCOMES:
Comparison of EVQ score to Timed Up and Go test | Day 0
  Timed Up and Go test (seconds)
Comparison of EVQ score to Timed Up and Go test | Month 1
  Timed Up and Go test (seconds)
Comparison of EVQ to unipedal stance test | Day 0
  Unipedal stance test (seconds)
Comparison of EVQ to unipedal stance test | Month 1
  Unipedal stance test (seconds)
Comparison of EVQ to Sternal Push Test | Day 0
  Sternal Push Test
Comparison of EVQ to Sternal Push Test | Month 1
  Sternal Push Test
Comparison of EVQ to Walking and talking test | Day 0
  Walking and talking test
Comparison of EVQ to Walking and talking test | Month 1
  Walking and talking test
Sensitivity of Balance and Daily Life Questionnaire to change | Month 1
  Balance and Daily Life Questionnaire given 30 days apart

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nimes, Nîmes, France

REFERENCES:
- [Result] De Labachelerie C, Viollet E, Alonso S, Dauvergne C, Blot M, Nouvel F, Fagart W, Chevallier T, Gelis A, Dupeyron A. Development and psychometric properties of the Balance in Daily Life (BDL) scale in a population of frail older people. Maturitas. 2024 Sep;187:108064. doi: 10.1016/j.maturitas.2024.108064. Epub 2024 Jul 8. PMID 39029351